CLINICAL TRIAL: NCT01279512
Title: Metformin vs. Acarbose Treatment in Infertile Overweight Women With PCOS: A Prospective Randomized Clinical Trial
Brief Title: Metformin Versus Acarbose Treatment in Infertile Overweight Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Royan-Emb-011
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2006-08

CONDITIONS: PCO
Keywords: Metformin Acarbose pco infertility overweight
MeSH Terms: interventions — Metformin; Acarbose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin reciepiants (Experimental): Infertile overweight women with PCO who received Metformin
  Interventions: Drug: Metformin
- Acarbose reciepiants (Experimental): Infertile overweight women with PCO who received Acarbose
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Metformin — The metformin dose will be 500 mg/ day in the first week, 1000 mg/ day in the second week and 1500 mg/ day for the next 10 weeks.
  Other Names: Metformin description
  Arms: Metformin reciepiants
Drug: Acarbose — Acarbose group will be treated by acarbose (its dose will be 100 mg/day in the first week, 200 mg/ day in the second week and 300 mg/ day for the next 10 weeks).
  Other Names: Acarbose description
  Arms: Acarbose reciepiants

SUMMARY:
This study is a prospective randomized clinical trial to compare the endocrine and metabolic effects of two anti diabetic drugs (metformin vs. acarbose) in infertile overweight women with PCOS

DETAILED DESCRIPTION:
This study is a prospective randomized clinical trial to compare the endocrine and metabolic effects of two anti diabetic drugs (metformin vs. acarbose) in infertile overweight women with PCOS.

Polycystic ovary syndrome (PCOS) is characterized by menstrual irregularity, hyperandrogenism, chronic anovulation and enlarged ovaries with more than twelve peripherally located follicles less than 10 mm in diameter. Hyperinsulinemia is one of the diagnostic features of PCOS and patients with PCOS are found to have resistance to either endogenous or exogenous insulin. Different insulin sensitizing drugs used for improvement of hyperinsulinemia in PCOS subjects. Metformin (N dimethyl-biguanide) is an anti diabetic drug that increases glucose utilization in insulin sensitive tissues. Acarbose is an alfa-Glycosidase inhibitor acts by slowing the absorption of carbohydrates from the intestine, prevents Glucosidase activity in the brush-border of the intestinal mucosa, decreasing disaccharide digestion, reducing enteric monosaccharide absorption, so minimizing the postprandial rise of blood glucose concentration. The aim of present study is to compare the endocrine and metabolic effects of these two antidiabetic drugs (metformin vs. acarbose) in infertile overweight women with PCOS.

The study population comprises all infertile patients with diagnosis of polycystic ovarian syndrome who were overweight (BMI>25Kg/m2). The PCO subjects will be recognized based on the Rotterdam criteria inclusive 1) irregular menstruation, 2) clinical and /or biochemical signs of hyperandrogenism, 3) polycystic ovaries (presence of 12 or more follicles in each ovary measuring 2-9 mm in diameter, and /or increased ovarian volume greater than 10 ml). Diagnosis of PCOS was confirmed by the presence two of three criteria beside the infertility.

In this study all eligible patients will be randomly allocated into two study groups by a computerized randomization method:

Acarbose group will be treated by acarbose (its dose will be 100 mg/day in the first week, 200 mg/ day in the second week and 300 mg/ day for the next 10 weeks). Metformin group will be received metformin. The metformin dose will be 500 mg/ day in the first week, 1000 mg/ day in the second week and 1500 mg/ day for the next 10 weeks.

Data collection will be performed by using questionnaire to be filled as per the available records and laboratory results. This study will be accomplished in Royan Institute on 50 PCO patients (25 patients in each group) and a continuous sampling method will be applied. Data analysis will be done through descriptive and perceptive statistical methods by using SPSS software version 15 for windows.

ELIGIBILITY:
Inclusion Criteria:

* Poly Cystic Ovarian Syndrome patients
* Age < 40 years
* BMI > 25 kg/m2

Exclusion Criteria:

* Smoking
* Overt diabetes mellitus, hyperprolactinemia, diseases that would disturb clinical and hormonal responses (adrenal disease or tumors, ovarian tumors, thyroid disease)
* The use of hormonal medications or drugs that might interfere with carbohydrate metabolism over the last 6 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Weight reduction (BMI improvement) | After 3 months of Metformin or Acarbose
  compare the effect of Metformin and Acarbose to weight reduction

SECONDARY OUTCOMES:
Fasting blood sugar (FBS) | two hours post prandial blood sugar
  Compare the effect of Metformin and acarbose to fasting blood sugar reduction
FSH | 6 months
  compare the effect of Metformin and Acarbose to decrease the level of FSH
LH | 6 months
  compare the effect of Metformin and Acarbose to decrease the level of LH
Estradiol | 6 months
  compare the effect of Metformin and Acarbose to decrease the Esteradiol level
Prolactin | 6 months
  compare the effect of Metformin and Acarbose to decrease the Prolactin level
Total testosterone | 6 months
  compare the the effect of Metformin and Acarbose to decrease Total testosterone level
Total cholesterol | 6 months
  comparethe the effect of Metformin and Acarbose to decrease total cholesterol level
triglyceride | 6 months
  comparethe the effect of Metformin and Acarbose to decrease the triglyceride level
High density Lipoprotein | 6 months
  compare the the effect of Metformin and Acarbose to decrease high density lipoprotein
Low density lipoprotein | 6 months
  compare the the effect of Metformin and Acarbose to decrease Low Density Lipoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Moini, MD, Study Chair — Scientific board; Elham Amirchaghmaghi, MD, Study Director — Invetigator; Zhila Ahmadi, BS.c, Principal Investigator — Investigator; Bita Eslami, MPH, Principal Investigator — Investigator; Ali asghar Akhlaghi, BS.c, Principal Investigator — Investigator; Reza salmanyazdi, MLD, Principal Investigator — Investigator
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: RoyanInstitute — http://www.royaninstitute.org